CLINICAL TRIAL: NCT00272636
Title: Randomized Comparison of Radiofrequency Catheter Ablation vs. Antiarrhythmic Therapy With Amiodarone for Maintaining Sinus Rhythm in Patients With Chronic Atrial Fibrillation
Brief Title: Radiofrequency Catheter Ablation for Chronic Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: San Raffaele University Hospital, Italy (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-0480
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2006-01

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; amiodarone; cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation; Amiodarone; Electric Countershock

INTERVENTIONS:
Procedure: Radiofrequency catheter ablation
Drug: Amiodarone and cardioversion

SUMMARY:
The purpose of this study is to determine the long-term efficacy of radiofrequency catheter ablation in patients with chronic atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic atrial fibrillation

Exclusion Criteria:

* Left atrial diameter >55 mm
* Left ventricular ejection fraction <0.30
* Contraindication to amiodarone therapy or anticoagulation with warfarin
* Presence of a mechanical prosthetic valve
* History of a cerebrovascular accident
* Presence of left atrial thrombus on TEE
* Prior attempt at catheter or surgical ablation for atrial fibrillation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2002-11; Study Completion 2005-02

PRIMARY OUTCOMES:
Freedom from atrial fibrillation and atrial flutter in the absence of antiarrhythmic drug therapy at 1 year.

SECONDARY OUTCOMES:
incidence of complications
changes in left atrial diameter
changes in left ventricular ejection fraction
changes in symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Oral, MD, Principal Investigator — University of Michigan; Fred Morady, MD, Study Chair — University of Michigan
Locations (2):
- University of Michigan Health System, Ann Arbor, Michigan, United States
- San Raffaele Hospital, Milan, Italy